CLINICAL TRIAL: NCT04980248
Title: A Phase 1, Open-label, Dose-escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ALXN1850 in Adults With Hypophosphatasia
Brief Title: Study of ALXN1850 in Participants With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN1850-HPP-101
Record Dates: First submitted 2021-07-23; First posted 2021-07-28 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Hypophosphatasia
Keywords: HPP; enzyme replacement therapy; low alkaline phosphatase; tissue-nonspecific alkaline phosphatase; TNSALP
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Intervention Model Description: Study participants will be enrolled into 3 cohorts in a sequential fashion.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN1850 (Experimental): Three experimental cohorts will be administered 3 dosages (low, medium, high) of ALXN1850, respectively, via IV infusion and/or SC over multiple administration intervals.
  Interventions: Biological: ALXN1850

INTERVENTIONS:
Biological: ALXN1850 — ALXN1850 will be administered as an IV infusion and via the SC route.

SUMMARY:
This is an open-label, dose-escalating study to assess safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and immunogenicity of ALXN1850 when given intravenous (IV) and subcutaneous (SC) to adults with HPP.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of HPP
* Not anticipated to require further treatment with enzyme replacement therapy to treat participant's HPP after study completion
* Willing and able to follow protocol-specified contraception requirements
* Willing and able to give informed consent

Exclusion Criteria:

* Primary or secondary hyperparathyroidism or hypoparathyroidism
* Fracture within 12 weeks of screening
* Current or relevant history of unstable physical or psychiatric illness
* Significant allergies
* Asfotase alfa use within 6 months and/or positive for asfotase alfa antidrug antibody/neutralizing antibodies

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Las Vegas, Nevada
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas

REFERENCES:
- [Derived] Dahir KM, Shannon A, Dunn D, Voegtli W, Dong Q, Hasan J, Pradhan R, Pelto R, Pan WJ. Safety, pharmacokinetics, and pharmacodynamics of efzimfotase alfa, a second-generation enzyme replacement therapy: phase 1, dose-escalation study in adults with hypophosphatasia. J Bone Miner Res. 2024 Sep 26;39(10):1412-1423. doi: 10.1093/jbmr/zjae128. PMID 39135540
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1850-HPP-101&attachmentIdentifier=8682c152-0932-4dfb-af33-423a6345591f&fileName=CSR_Synopsis_alxn1850hpp101_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Participants received 15 milligrams (mg) of ALXN1850 as a single intravenous dose, followed by 15 mg of ALXN1850 as a subcutaneous injection at 1-week interval for 3 doses.
- Cohort 2: Participants received 45 mg of ALXN1850 as a single intravenous dose, followed by 45 mg of ALXN1850 as a subcutaneous injection at 1-week interval for 3 doses.
- Cohort 3: Participants received 90 mg of ALXN1850 as a single intravenous dose, followed by 90 mg of ALXN1850 as a subcutaneous injection at 1-week interval for 3 doses.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 5 | 5 | 5
Received at Least 1 Dose of Study Drug | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received any amount of study drug. Participants were analyzed according to the study drug received.
Groups:
- Cohort 1: Participants received 15 mg of ALXN1850 as a single intravenous dose, followed by 15 mg of ALXN1850 as a subcutaneous injection at 1-week interval for 3 doses.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.44) | 37.8 (12.52) | 54.6 (9.07) | 45.5 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 11
  Male | 2 | 2 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: TEAEs were defined as any adverse events (AEs) that began or worsened on or after the first dose of treatment until the final follow-up visit. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. TESAEs were defined as any serious AEs that began or worsened on or after the first dose of treatment until the final follow-up visit. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 up to Day 85
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Participants received 15 mg as a single intravenous dose, followed by 15 mg subcutaneous at 1-week interval for 3 doses.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Participants
  TEAEs | 3 | 5 | 4
  TESAEs | 0 | 0 | 1

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of ALXN1850 Following Intravenous (IV) Dose, Subcutaneous (SC) Dose 1, SC Dose 2 and SC Dose 3
Time Frame: Predose, 2, 6 and 12 hours postdose on Days 1, 15, 22 and 29
Population: The Pharmacokinetic (PK) Set included all treated participants for whom the PK profile of ALXN1850 was adequately characterized. PK analyses was based upon the study drug received. Here, number analyzed signifies those participants who were evaluable for prespecified categories only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
micrograms/milliliter
  IV Dose | 5.31 (29.2) | 13.5 (23.3) | 32.4 (31.1)
  SC Dose 1 | 0.871 (43.8) | 2.89 (59.4) | 8.60 (43.5)
  SC Dose 2: number analyzed (Participants) | 5 | 4 | 5
  SC Dose 2 | 0.815 (52.3) | 2.38 (88.8) | 6.33 (55.5)
  SC Dose 3: number analyzed (Participants) | 5 | 4 | 4
  SC Dose 3 | 0.844 (75.2) | 2.41 (97.4) | 5.44 (145)

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity Following IV Dose of ALXN1850
Time Frame: Predose, 2, 6 and 12 hours postdose on Days 1, 15, 22 and 29
Population: The PK Set included all treated participants for whom the PK profile of ALXN1850 was adequately characterized. PK analyses was based upon the study drug received. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms/milliliter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
hour*micrograms/milliliter | 407 (38.3) | 1010 (26.0) | 2450 (33.6)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Dosing Interval (AUCtau) Following SC Dose 1, SC Dose 2 and SC Dose 3
Time Frame: Predose, 2, 6 and 12 hour postdose on Days 1, 15, 22 and 29
Population: The PK Set included all treated participants for whom the PK profile of ALXN1850 was adequately characterized. PK analyses was based upon the study drug received. Here, overall number of participants analyzed signfies those participants who were evaluable for this endpoint only and number analyzed signifies those participants who were evaluable for prespecified categories only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms/milliliter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 4
hour*micrograms/milliliter
  SC Dose 1 | 115 (42.2) | 383 (58.1) | 1110 (49.6)
  SC Dose 2: number analyzed (Participants) | 5 | 4 | 4
  SC Dose 2 | 111 (58.5) | 350 (83.3) | 872 (65.5)
  SC Dose 3: number analyzed (Participants) | 5 | 4 | 4
  SC Dose 3 | 115 (73.9) | 367 (95.6) | 881 (104)

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Dosing Interval (AUCtau) Values of the First SC Versus IV Administration of ALXN1850
Time Frame: Predose, 2, 6 and 12 hour postdose on Days 1, 15, 22 and 29
Population: The PK Set included all treated participants for whom the PK profile of ALXN1850 was adequately characterized. PK analyses was based upon the study drug received. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure only. As pre-specified, data are presented pooled for all participants who received study drug.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Groups:
- All Participants: Participants received 15, 45 or 90 mg of ALXN1850 as a single intravenous dose, followed by 15, 45 or 90 mg of ALXN1850 as a subcutaneous injection at 1-week interval for 3 doses.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Ratio
  15 mg | 0.286 [0.105 to 0.782]
  45 mg | 0.367 [0.180 to 0.784]
  90 mg | 0.368 [0.0908 to 1.49]

6. Secondary Outcome: Absolute Change From Baseline in Plasma Concentration of Pyridoxal-5' Phosphate (PLP) at Week 1
Time Frame: Baseline, 1 Week post Day 1 IV dose and 1 Week post Day 29 SC dose 3
Population: The Pharmacodynamic (PD) Set included all treated participants for whom the PD profile of ALXN1850 was adequately characterized. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure only. Here, number analyzed signifies those participants who were evaluable for prespecified timepoints only.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
nanogram/milliliter
  1 Week post Day 1 IV Dose: number analyzed (Participants) | 1 | 1 | 1
  1 Week post Day 1 IV Dose | -18.300 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -7.600 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -49.460 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant.
  1 Week post Day 29 SC Dose 3 | -97.950 (164.0193) | -38.573 (26.4932) | -28.055 (17.3237)

7. Secondary Outcome: Absolute Change From Baseline in Plasma Concentration of Inorganic Pyrophosphate (PPi) at Week 1
Time Frame: Baseline, 1 Week post Day 1 IV dose and 1 Week post Day 29 SC dose 3
Population: The PD Set included all treated participants for whom the PD profile of ALXN1850 was adequately characterized. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure only. Number analyzed signifies those participants who were evaluable for the prespecified timepoints only.
Measure: Mean (Standard Deviation); unit: micromoles (uM)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 1
micromoles (uM)
  1 Week post Day 1 IV Dose: number analyzed (Participants) | 1 | 1 | 0
  1 Week post Day 1 IV Dose | -1.620 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -1.930 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. |
  1 Week post Day 29 SC Dose 3 | -0.813 (0.5970) | -1.505 (0.1202) | -2.040 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant.

8. Secondary Outcome: Absolute Change From Baseline in Plasma Concentration of Pyridoxal Phosphate/ Pyridoxal (PLP/PL) Ratio at Week 1
Time Frame: Baseline, 1 Week post Day 1 IV dose and 1 Week post Day 29 SC dose 3
Population: The PD Set included all treated participants for whom the PD profile of ALXN1850 was adequately characterized. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure only. Here, number analyzed signifies those participants who were evaluable for prespecified timepoints only.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
Ratio
  1 Week post Day 1 IV Dose: number analyzed (Participants) | 1 | 1 | 1
  1 Week post Day 1 IV Dose | -8.570 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -16.070 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -15.260 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant.
  1 Week post Day 29 SC Dose 3 | -7.620 (5.3878) | -15.285 (6.2807) | -8.368 (6.3951)

9. Secondary Outcome: Percent Change From Baseline in Plasma Concentration of PLP at Week 1
Time Frame: Baseline, 1 Week post Day 1 IV dose and 1 Week post Day 29 SC dose 3
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
percent change
  1 Week post Day 1 IV Dose: number analyzed (Participants) | 1 | 1 | 1
  1 Week post Day 1 IV Dose | -47.906 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -17.512 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -86.318 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant.
  1 Week post Day 29 SC Dose 3 | -33.895 (42.5254) | -69.049 (16.5385) | -70.515 (23.0447)

10. Secondary Outcome: Percent Change From Baseline in Plasma Concentration of PPi at Week 1
Time Frame: Baseline, 1 Week post Day 1 IV dose and 1 Week post Day 29 SC dose 3
Population: The PD Set included all treated participants for whom the PD profile of ALXN1850 was adequately characterized. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure only. Number analyzed signifies those participants who were evaluable for prespecified timepoints only.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 1
percent change
  1 Week post Day 1 IV Dose: number analyzed (Participants) | 1 | 1 | 0
  1 Week post Day 1 IV Dose | -53.821 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -70.956 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. |
  1 Week post Day 29 SC Dose 3 | -32.740 (23.0615) | -55.328 (1.7622) | -71.329 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant.

11. Secondary Outcome: Percent Change From Baseline in Plasma Concentration of PLP/PL Ratio Over Time at Week 1
Time Frame: Baseline, 1 Week post Day 1 IV dose and 1 Week post Day 29 SC dose 3
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
percent change
  1 Week post Day 1 IV Dose: number analyzed (Participants) | 1 | 1 | 1
  1 Week post Day 1 IV Dose | -65.270 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -92.944 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant. | -91.323 (NA) — Standard deviation could not be calculated as there was only 1 evaluable participant.
  1 Week post Day 29 SC Dose 3 | -35.104 (15.0384) | -77.160 (16.0636) | -60.816 (49.7578)

12. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Positive and Neutralizing Antibody (NAb) Positive Status
Time Frame: Baseline up to Day 85
Population: The Immunogenicity Analysis Set included all treated participants who received any study drug and who after the first dose had at least one reportable result in the ADA assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Participants
  ADA Positive | 2 | 0 | 2
  NAb Positive | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 85
Description: All-cause mortality is reported for all enrolled participants. Serious adverse events and other adverse events are reported in the Safety Set, which included all participants who received any amount of study drug. Participants were analyzed according to the study drug received.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 3/5 | 5/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=5) | Cohort 3 (N=5)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=5) | Cohort 3 (N=5)
Fatigue (General disorders) | 1 | 1 | 0
Injection site bruising (General disorders) | 1 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 1
Injection site haemorrhage (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Dizziness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0/3 | 0/3 | 1 — This AE is gender specific. So, the number of participants at risk is the female population only.
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Abdominal pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Nausea (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Hyperphosphaturia (Renal and urinary disorders) | 0 | 1 | 0
Dry eye (Cardiac disorders) | 0 | 1 | 0
Breast discomfort (Reproductive system and breast disorders) | 0/3 | 0/3 | 1 — This AE is gender specific. So. the number of participants at risk is the female population only.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT04980248/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT04980248/SAP_001.pdf